CLINICAL TRIAL: NCT02250456
Title: Detect, Monitor and Prevent Vascular Abnormalities Associated With Turner Syndrome
Brief Title: AVAST Anomalies Vasculaires Associées au Syndrome de Turner (Vascular Abnormalities Associated With Turner Syndrome)
Acronym: AVAST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5545
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Turner Syndrome; Peripheral Angiopathy; Vascular Malformation; Lymphedema
MeSH Terms: conditions — Turner Syndrome; Peripheral Vascular Diseases; Vascular Malformations; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Turner syndrome patients and vascular abnormalities
  Interventions: Procedure: Echo doppler

INTERVENTIONS:
Procedure: Echo doppler — vascular ultrasound explorations

SUMMARY:
Turner syndrome is a genetic condition, rare, due to the total or partial absence of one X chromosome, affecting 1/2500 newborn female. It combines almost constantly short stature and ovarian failure with infertility.

Other anomalies are inconstant: morphological characteristics of varying intensity, associated malformations, and increased risk of acquired diseases ...

The prognosis of patients reaching the Turner Syndrome is linked to cardiovascular complications (congenital heart disease, dilatation of the ascending aorta with risk of dissection or rupture of aneurysm), causing early mortality with reduction of life expectancy of at least 10 years.

For these reasons, screening for heart disease and dilatation of the ascending aorta is established and is intended to prevent the complications associated with medical treatment and / or surgery to increase life expectancy and reduce the co-morbidities.

On the vascular level, the recommendations other than those relating to the monitoring of the diameter of the ascending aorta include research of renal artery stenosis by doppler ultrasound if the patient is hypertensive and looking for lymphedema.

However, other arterial lesions were described in the literature, outside of the aneurysm of the ascending aorta. These peripheral arterial lesions can also be life and / or functional prognosis of the patient. Ascending aorta dilation seems not to be exclusive in Turner syndrome.

In addition, specific vascular lesions outside the affected artery are described: hepatic cirrhosis by vascular depletion, lymphedema and varicose veins. The prevalence of venous or lymphatic disease is unknown.

A single-center review of 9 cases of patients followed at the University Hospital of Strasbourg showed the presence of vascular lesions discovered incidentally during assessments performed for reasons other than cardiovascular screening: cystic lymphangioma, internal carotid aneurysm, agenesis of the inferior vena cava, early varicose veins, embryonic cerebral artery, etc ... None of these patients showed any dilatation of the ascending aorta or heart disease. Peripheral vascular abnormalities in this patient group are exclusive.

In this study, we seek to demonstrate that arterial disease in Turner syndrome involve the entire arterial territory and is not confined to the ascending aorta. Screening for arterial lesions should be performed on the entire arterial vascular tree and regularly in the course of time, especially as the presence of cardiovascular risk factors increases with the age of these patients.

The venous and lymphatic vascular damage in the literature and in our series of cases in University Hospital of Strasbourg description should also lead to the detection of these lesions.

These vascular complications can be alone responsible for the reduction in life expectancy or responsible for serious morbidity. Improved screening of associated vascular lesions is necessary to enable the best prevention of cardiovascular complications.

It is also to establish the prevalence of vascular anomalies, whether arterial, venous or lymphatic, to better understand the disease and its management. By collecting systematically karyotype leading to diagnosis, it may be possible to make a link between the genetic defect and heart or vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Any woman over 18 years with Turner Syndrome confirmed by karyotype
* Affiliated to a social security scheme
* Having signed an informed consent
* Having been informed of the results of the medical examination prior

Exclusion Criteria:

* Inability to give informed patient information related to comprehension difficulties
* Topic featuring against-indications for MRI examination:

  * pacemaker or automatic defibrillator, implanted pump
  * auditory nerve stimulator, anal nerve stimulator, etc ...
  * the ferromagnetic objects in the soft tissues, intraocular metallic objects, cerebral vascular clips
  * claustrophobia
  * morphotype not allowing access to MRI
* Patient under judicial protection, guardianship or trusteeship
* Patient in exclusion period (as determined by a previous study or in progress)
* Pregnancy at the time of inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with Turner Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical events and systematized vascular ultrasound explorations | Annual evaluation with a 5 years follow-up
  Reports of annual clinical events and results of complementary cardiovascular investigations.
  Systematized arterial and venous ultrasound explorations once a year. Reports karyotype used to put the diagnosis of turner Syndrome to perform correlations karyotype - phenotype and karyotype - event.
  Annual standardized biological exploration.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GAERTNER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (6):
- France (6):
  - Service de Chirurgie et Médecine Vasculaire, CHU Jean Minjoz, Besançon
  - Service d'Angiologie, CHU Bocage, Dijon
  - Service de gynécologie, Centre Médico Chirurgical Obstétrical, Hôpitaux Universitaires, Schiltigheim
  - Service d'endocrinologie, Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service d'explorations fonctionnelles non invasives cardio-vasculaires, Nouvel Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service HTA, maladies vasculaires et pharmacologie clinique, Nouvel Hôpital Civil, Hôpitaux Universitaires, Strasbourg